CLINICAL TRIAL: NCT07324083
Title: Immediate Implant Loading Following Ridge Preservation: A Randomized Controlled Trial Comparing Autogenous Mineralized Dentin Graft and Beta-Tricalcium Phosphate
Brief Title: Immediate Implant Loading After Ridge Preservation Using Autogenous Dentin Graft and Beta-Tricalcium Phosphate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soaad Tolba Mohammed Tolba Badawi (Other)
Responsible Party: Sponsor-Investigator, Soaad Tolba Mohammed Tolba Badawi, Lecturer of Oral and Maxillofacial Surgery, Faculty of Dentistry, Mansoura University, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.25.12.95
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Tooth Extraction; Alveolar Ridge Preservation; Immediate Implant Loading
Keywords: Socket preservation; immediate loading; autogenous dentin graft; beta-tricalcium phosphate; dental implant
MeSH Terms: interventions — beta-tricalcium phosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autogenous Mineralized Dentin Graft (Active Comparator): Extraction sockets were preserved using AMDG prepared from the patient's own extracted tooth. Implants were placed 6 months post-grafting and immediately loaded within 48 hours.
  Interventions: Procedure: Autogenous Mineralized Dentin Graft
- Beta-Tricalcium Phosphate (Active Comparator): Extraction sockets were preserved using synthetic β-TCP bone graft. Implants were placed 6 months post-grafting and immediately loaded within 48 hours.
  Interventions: Procedure: Beta-Tricalcium Phosphate
- Control (Ungrafted Socket) (Placebo Comparator): Extraction sockets were left ungrafted and allowed to heal naturally. Implants were placed 6 months post-extraction and immediately loaded within 48 hours.
  Interventions: Procedure: Control (Ungrafted Socket)

INTERVENTIONS:
Procedure: Autogenous Mineralized Dentin Graft — Extraction sockets were preserved using AMDG prepared from the patient's own extracted tooth. Implants were placed 6 months post-grafting and immediately loaded within 48 hours.
  Arms: Autogenous Mineralized Dentin Graft
Procedure: Beta-Tricalcium Phosphate — Extraction sockets were preserved using synthetic β-TCP bone graft. Implants were placed 6 months post-grafting and immediately loaded within 48 hours.
  Arms: Beta-Tricalcium Phosphate
Procedure: Control (Ungrafted Socket) — Extraction sockets were left ungrafted and allowed to heal naturally. Implants were placed 6 months post-extraction and immediately loaded within 48 hours.
  Arms: Control (Ungrafted Socket)

SUMMARY:
This randomized controlled clinical trial aimed to evaluate the clinical, radiographic, and histological outcomes of immediate implant loading in extraction sockets preserved using autogenous mineralized dentin graft (AMDG), beta-tricalcium phosphate (β-TCP), or no grafting. Twenty-two patients requiring extraction of maxillary premolars were enrolled, contributing a total of 27 extraction sites. Sites were randomly allocated into three groups: AMDG, β-TCP, or ungrafted control.

Following socket preservation, dental implants were placed after a 6-month healing period and immediately loaded within 48 hours. Alveolar ridge dimensional changes were assessed using cone-beam computed tomography (CBCT) between implant placement and 2 years post-loading. Implant stability, peri-implant soft tissue health, and probing depths were evaluated at loading and during follow-up visits. Histological evaluation of regenerated bone was performed at the time of implant placement.

The study sought to determine whether AMDG provides comparable or superior outcomes to β-TCP and ungrafted sockets in supporting immediate implant loading.

DETAILED DESCRIPTION:
Immediate implant loading requires adequate primary stability and sufficient bone volume and quality. Ridge preservation techniques are therefore critical in maintaining post-extraction socket dimensions. Autogenous dentin grafts have recently gained attention due to their osteoconductive properties, biocompatibility, and cost-effectiveness.

This study compares AMDG with a commonly used synthetic graft material (β-TCP) and ungrafted sockets to assess their influence on ridge preservation, implant stability, peri-implant tissue health, and bone quality under immediate loading conditions.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older
* Patients requiring extraction of a maxillary premolar tooth
* Adequate bone height to allow delayed implant placement
* Good oral hygiene and compliance with follow-up visits
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria

* Presence of uncontrolled systemic diseases that could affect bone healing
* History of radiotherapy to the head and neck region
* Heavy smoking
* Active infection or untreated periodontal disease at the extraction site
* History of bisphosphonate or other antiresorptive drug use
* Poor oral hygiene or inability to comply with study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Alveolar Ridge Width Change | From 6 months post-extraction (implant placement) to 2 years post-loading
  Dimensional changes in alveolar ridge width were assessed using CBCT at the center, mesial, and distal sections of each implant site. Measurements were compared between the grafted (AMDG and β-TCP) and control groups over the follow-up period.Unit of Measure: Millimeters (mm)

SECONDARY OUTCOMES:
Implant Stability Quotient (ISQ) | At implant loading, 3 months, and 6 months post-loading
  Implant stability was assessed using resonance frequency analysis to record ISQ values at each follow-up visit for all groups.Unit of Measure: ISQ units(0-100)
Modified Sulcus Bleeding Index (mSBI) | At implant loading, 3 months, and 6 months post-loading
  Peri-implant soft tissue inflammation was evaluated using the mSBI at each follow-up visit for all groups. Unit of Measure: Index score (0-5 scale)
Probing Pocket Depth (PPD) | At implant loading, 3 months, and 6 months post-loading
  Probing depth around each implant was measured using a periodontal probe to assess peri-implant tissue health across all groups.Unit of Measure: Millimeters (mm)
Histological Bone Quality | 6 months post-grafting (at implant placement)
  Histological analysis of bone biopsies obtained from grafted and control sites was performed to evaluate bone maturity, remodeling, and osseointegration. Unit of Measure: Qualitative histological score.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided